CLINICAL TRIAL: NCT05104385
Title: Hacettepe Health Cohort: A Prospective Follow-up of the General Health Status and Effectiveness, Durability and Adverse Effects of COVID-19 Vaccine Among Students of Medical and Dental Schools
Brief Title: Hacettepe University COVID-19 Vaccinated's Health Cohort- Students of Health Sciences
Acronym: HU-CoVaCS
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Banu Cakir, Principal Investigator, Hacettepe University
Other Study IDs: TCP-2021-19467
Record Dates: First submitted 2021-10-31; First posted 2021-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pandemic; SARS-CoV2 Infection; Immunization; Infection; Health
Keywords: COVID-19; vaccine-induced immunity; CoronaVac- inactivated vaccine; Biontech- mRNA vaccine; prospective cohort; health personnel
MeSH Terms: conditions — COVID-19; Infections | interventions — Longitudinal Studies; RNA, Messenger; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples are drawn, at fasting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hacettepe University Health Cohort- Students of Health Sciences: Students of medical school (grades 4,5, and 6) in 2021 Spring Students of dental school (grades 4 and 5) in 2021 Spring New comers of grade 4 in both medical and dental school will be recruited early in October 2021.
  There is no intervention. Vaccinations for COVID-19 have been provided by the Turkish Ministry of Health, in a pre-planned schedule. The study will follow students after vaccination, regardless of the type and dose administered.
  Interventions: Other: Observational, prospective, follow-up of the recipients of CoronaVac (inactivated), Pfizer-Biontech (mRNA) vaccines

INTERVENTIONS:
Other: Observational, prospective, follow-up of the recipients of CoronaVac (inactivated), Pfizer-Biontech (mRNA) vaccines — Based on the Turkish Ministry of Health regulations, any research protocol involving use of any drug/vaccine needs to be presented in a clinical trial format, and is presented to the clinical research ethical boards accordingly. Otherwise, the study has no intervention (to the exposure status) involved. Selection, administration, number of doses applied and the period between vaccine doses are beyond the capacity the study team.

SUMMARY:
The first COVID-19 case in Turkey was reported on March 11, 2000. National COVID-19 mass vaccination was initiated on Jan 13, 202, with two doses of CoronaVac (R) inactivated vaccine (of Sinovac), 28 days apart. The health personnel were prioritized in the mass vaccination, given their high rates of exposure and fatality. National COVID-19 statistics have been limited to those announced in the media; data breakdown by gender, age, vaccine type and status etc. is not provided, nor is the association between non-pharmaceutical preventive measures (NPPM) and infection rates. Well-planned, longitudinal, detailed studies with laboratory support are clearly warranted. Hacettepe University is a leading institution in Turkey, with its large health sciences campus. Students of medical school (grades 4, 5, and 6) and dental school (grades 4 and 5) have been actively providing patient care in HU Hospitals, and more than 10% of medical interns had been reportedly diagnosed as COVID-19 cases prior to vaccination activities, despite (reportedly) strict non-pharmaceutical public preventive measures (NPPM) use inside/outside the occupational settings. A two-year prospective cohort study was planned for periodic evaluation of students' general health status and COVID-19 risk/exposure/infection, for timely referrals and quarantine/isolation, as needed. Anti- SARS-CoV-2-RBS antibodies will be measured periodically after vaccination, together with evaluation of potential adverse effects, presence and durability of vaccine-induced immunity. Comparison of antibody levels were planned for incident COVID-19 cases and two test-negative controls of the same gender, attending the same grade and faculty. A subcohort will be followed for aymptomatic infection risk. Institutional ethical approvals were obtained, as required. A step-wise informed consent was obtained from all participants, all tests will be done with de-personalized records, and all statistical analyses and reporting will be completed anonymously. Follow-up of participants will be ensured using participant-specific study identification numbers provided at enrollment. Study team is composed of academic personnel of 10 selected departments, nursing support is provided by the Students' Health Center in the Campus, and dental faculty are assigned for obtaining informed during the 4 subsequent study visits. The budget of the study is provided by the Hacettepe University Scientific Research Projects Office (BAP).

DETAILED DESCRIPTION:
The study was planned, and ethical approval procedures were initiated in late January, 2021. However, serial official approval processes delayed the initiation of the study beyond the pre-planned initiation date (late in March 2021, to catch the 28th day after the second dose of CoronaVac vaccine). Thus, the study plan was revised, and so were the approval processes.

The planned prospective cohort study started its recruitment process in June, with the first enrollment on June 21, 2021. The study is an open cohort; vaccination times vary, some students participated in the first visit, but have/can leave the study before May 2023 (the planned closure time for testing); some students did not participate in the first visit (in June-July 2021), yet preferred to be involved in the study bythe time of the second visit (October 2021) and so.

Participants are being recruited from students of medical school (grades 4,5, and 6) and dental school (grade 4 and %), and are involved in the study for all/some of the procedures offered. The study aimed to:

1. Investigate the sociodemographic characteristics, health status, life habits, quality of life (via validated indices), COVID-19 status, vaccination status for SARS-CoV-2, use of non-pharmaceutical preventive measures against COVID-19. These will be accomplished through online, depersonalized, self-completed standardized questionnaire and use of validated scales.;
2. Complete anthropometric measures and physical examination at each visit;
3. Check blood levels for complete blood count, renal function tests, liver enzymes, D-dimer, vitamin D, HbA1c levels, and lipid profile;
4. Check vaccine-induced immunity using quantitative, Anti-SARS-CoV-2 Receptor Binding Domain kit (Abbott Laboratories) at enrolment and each subsequent visits;
5. Evaluate the durability of vaccine-induced immunity, as measured by antibody levels periodically (at 3rd, 6th, 12th and 24th month after full immunization following full vaccination, i.e. 2 doses plus 28 days);
6. The cohort will be followed up to 24 months (through September 2023) for detecting COVID-19 infection and/or related hospitalization, intensive care unit (ICU)-admission or death; also, to study the potential association with personal risk factors and/or vaccine-induced immunity;
7. A nested, test-negative case-control study is integrated into the the cohort, such that each time a new COVID-19 case is identified (with a PCR-positivity), two gender and school/grade matched controls will be invited for PCR testing. Blood will be drawn from PCR test negative controls at the day (or within 1 day later) of the PCR-positivity of the case detected. This nested case-(test-negative) control design will enable to study the association between infection and current Anti-Spike1 RBD antibody levels, controlling for personal risk factors;
8. Given the considerable amount of asymptomatic infections among vaccinated individuals, 150 participants will be selected from among volunteers for 6 consecutive PCR-testing, with 15 days intervals between each testing.

Three study designs will be used to reach study objectives; namely, a large prospective cohort (for evaluating changes in general health status and neutralizing antibody levels, as measured by SARS-CoV-2-RBD Abs); a subcohort for periodical PCR testing to detect asymptomatic infection rates;

Over the course of the planned study, Pfizer-Biontech (R) m-RNA vaccination has been introduced for mass vaccination, as 2 doses, 28 days apart. Also, the Ministry of Health promoted a third dose of COVID-19 vaccination for health personnel in particular, due to rapidly decreasing immunity for COVID-19 among 2-dose CoronaVac vaccinated individuals. This change in mass vaccination introduced variation in our exposure status. Accordingly, the objectives of the study extended to calculation and comparison of the incidence-rates of COVID-19 infection and related complications among those vaccinated with either of the 2 vaccines (namely, CoronaVac and Biontech), controlling for the first doses and boosters, including mix-and-matches.

The four visits of the main cohort was completed as of July 7, 2023 (as planned). Preliminary findings have been published in a Turkish peer-reviewed medical journal. Due to administrative issues, periodic PCR-based asymptomatic case detection was postponed- will be resumed in Fall 2023 (if case numbers increase). The nested case-control sub-study will continue through November 1, 2023, as PCR-confirmed cases appear. So far, we have a total of 194 cases since the initiation of the cohort; 154 of these were detected by the cohort team, others were detected outside the cohort facility, but all were confirmed (upon students' approval) through personal electronic health records. The study is anticipated to finish by december 7, 2023. The unexpected 3 months of delay at initiation of the study (due to the time lag for the ethical approval process at the Ministry of Health) led to an expansion in data analysis and final reporting of the study (registered as December 7, 2023, by the University Scientific Research Unit, which is the sole funder of the study.)

ELIGIBILITY:
Inclusion Criteria:

1) students of the medical school (grades 4,5 and 6) in 2021 Spring semester 2 )students of the dental school (grades 4 and 5) in 2021 Spring semester 3) new comers of grade 4 of medical and dental school in 2021 Fall semester 4) those providing informed consent to participate in the study.

Exclusion Criteria:

None.

Ages: 20 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population is a sample of senior students of Hacettepe University medical and dental students, who actively work in Hacettepe hospitals during COVID-19 pandemic and, thus, have the potential for contacting COVID-19 infected individuals.
  The study team will approach all eligible students. Yet, participation in the study is totally voluntary, thus, the final sample is not expected to be a random sample of all eligibles.
  Study participants will be motivated to be in the study through graduation or study completion date, which ever come earlier.
Sampling Method: Non-Probability Sample
Enrollment: 1223 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Vaccine-induced immunity (status and durability) against SARS-CoV-2 | 21 June 2021-7 July 2023
  Anti-SARS-CoV-2 Spike 1 RBD antibodies are measured as a surrogate measure for vaccine-induced immunity
General health status (physical, mental, social) | 21 June 2021-7 July 2023
  Status and change in the self-reported morbidity and validated scales-based mental health status and quality of life will be followed over time.

SECONDARY OUTCOMES:
COVID-19 infection and related health complications | 21 June 2021-7 December 2023
  Incident cases of PCR-test positive COVID-19 cases, related hospitalization, intensive care unit (ICU) stay and death

CONTACTS AND LOCATIONS:
Overall Officials: Banu Cakir, Study Director — Hacettepe University, Division of Epidemiology (Chair)
Locations (1):
- Hacettepe University, Sıhhiye Campus, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All steps of the study have been completed using depersonalized data, based on participant-specific study code numbers provided at baseline visit. Individual participant data have been shared by the core study team members (n=3) only. Tabulated data have been shared with other researchers. Anonymized data have been saved for future enquiries (e.g., manuscripts, etc): Only three core team members (including principal investigator) have access to participant IDs and corresponding personal characteristics (including the national ID number).

REFERENCES:
- [Background] E. Karadogan Et Al. ,
- See also: paper publisher in a peer-reviewed journal, in Turkish — https://www.klimikdergisi.org/tr/2023/03/06/hacettepe-universitesi-saglik-ve-covid-19-kohortu/
- See also: indexed in Turkish scientific index — https://search.trdizin.gov.tr/tr/yayin/detay/1167355/hacettepe-saglik-kohortu-hu-covacs-calisma-tasarimi-baslangic-viziti-degerlendirmesi-ve-covid-19-asililarin-ilk-uc-aylik-takip-verileri